CLINICAL TRIAL: NCT07057310
Title: Aging Well: Targeting Obesity With GLP-1 Agonists to Enhance Physical and Vascular Health in Postmenopausal Women
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maria Daniela Hurtado Andrade, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-010834
Record Dates: First submitted 2025-05-05; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Menopause
Keywords: obesity; vascular function; aging; postmenopause; women
MeSH Terms: conditions — Obesity | interventions — semaglutide; Tirzepatide

STUDY DESIGN:
Intervention Model Description: This will be a 24-week, open-label, pragmatic, randomized clinical trial. Participants will be randomized 1:1 to receive tirzepatide or semaglutide with a standard lifestyle intervention or a lifestyle intervention alone. Tirzepatide or semaglutide will be started at the lowest dose and titrated every four weeks, as tolerated, up to the maximum dose of 2.4 mg weekly for semaglutide and 15 mg weekly for tirzepatide. The choice of the medication will depend on patient's preference, cost, and drug availability. We will assess body composition, measurements of physical function, obtain a blood sample for the measurement of aging biomarkers, and perform vascular testing at different timepoints.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight loss medication and standard lifestyle intervention (Experimental): Subjects will receive tirzepatide or semaglutide in combination with a standard lifestyle intervention.
  Interventions: Drug: semaglutide or tirzepatide; Behavioral: Lifestyle modification intervention
- Standard lifestyle intervention only (Active Comparator): Subjects will receive standard of care lifestyle intervention only.
  Interventions: Behavioral: Lifestyle modification intervention

INTERVENTIONS:
Drug: semaglutide or tirzepatide — Semaglutide and tirzepatide will be dosed as per prescription labels
  Arms: Weight loss medication and standard lifestyle intervention
Behavioral: Lifestyle modification intervention — All participants will be recommended the following: 1) low-calorie diet based on their predicted by Harris Benedict resting energy expenditure minus 500 kcal per day; 2) physical activity: a goal of 10,000 steps or more per day; 3) exercise: a goal of 150 minutes or more of moderate-intensity aerobic activity (cardiovascular exercise) per week; 4) limited consumption of liquid calories (i.e. sodas, juices, alcohol, etc.).

SUMMARY:
In postmenopausal women, obesity increases the risk of physical function decline, premature aging, and vascular dysfunction. Semaglutide and tirzepatide are potent obesity medications. The goal is to determine the effect of weight loss induced by the new generation of GLP-1 receptor agonists on physical function, aging biomarkers, and vascular function in postmenopausal women with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (with menopause defined as the cessation of menstrual periods for at least 12 months or history of bilateral oophorecomy)
* Age 46-60 years old
* BMI ≥ 30 kg/m2.

Exclusion Criteria:

* Past or current use of menopausal hormone therapy
* Early or premature menopause
* History of chemically induced menopause
* Impaired renal function (GFR ≤29)
* Thyroid-stimulating hormone ≥7 with low free T4
* Diabetes
* Cardiovascular disease
* Elevated blood pressure (>170/>95)
* Uncontrolled co-morbidities including inflammatory, autoimmune, infectious, hepatic, gastrointestinal, malignant, or psychiatric disease
* >5% change in weight during the 3 months prior to screening
* Other anti-obesity medication use within the past 3 months
* History of bariatric surgery
* History of malignant neoplasms within the past 5 years prior to screening
* Current use of supplements known to affect weight
* Personal or family history of medullary thyroid cancer.
* Wheelchair bound
* Vision loss

Ages: 46 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Cis-Gender
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Physical Function Measure: Short Physical Performance Battery (SPPB) score. | 24 weeks
  The SPPB is a standardized test that evaluates lower extremity function using three components: balance tests (standing in various positions), gait speed (walking a short distance), and chair stand (repeated standing from a seated position). Each component is scored from 0 to 4; the total score ranges from 0 to 12. Higher scores represent better physical function.
Physical Function Measure: Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) performed on the Rehabilitation Artificial Physical Intelligence Database (RAPID) foot pressure mat | 24 weeks
  The mCTSIB assesses balance under four sensory conditions: eyes open/closed on firm and foam surfaces. Testing is performed while standing on the RAPID foot pressure mat, which captures center of pressure and postural sway data. The primary measure is average sway area of the four sensory conditions. The sway area is the area which is required to correct equilibrium, representing the total area covered by postural sway, measured in square centimeters (cm²).
Physical Function Measure: Standing Chest Throw Test with a 2-kg Weighted Ball using Motion Sensor Technology (MST) | 24 weeks
  This test evaluates upper body muscular power. Participants perform a two-handed chest throw of a 2-kg medicine ball from a standing position. The MST is used to record throw distance, velocity, and related performance metrics. The primary measure is Peak Power Score (W).
Physical Function Measure: Chair-to-Stand Tests using Motion Sensor Technology (MST) | 24 weeks
  This test assesses lower body strength and function. Participants are instructed to stand up from a chair and sit back down five times without using their arms. The MST measures movement dynamics. The primary measure is peak power score (W).
Physical Function Measure: Six-Minute Walk Test (6MWT) | 24 weeks
  The 6MWT is a standardized submaximal exercise test used to assess functional aerobic capacity. Participants are instructed to walk as far as possible in six minutes along a flat, straight course. The total distance walked is recorded in feet. Longer walking distances indicate better aerobic capacity and endurance.
Physical Function Measure: Hand Grip Strength using a Hydraulic Hand Dynamometer | 24 weeks
  Participants are instructed to squeeze the dynamometer with maximum effort, measured in kilograms. The highest value from multiple trials is recorded.
Physical Function Measure: Short Form-12 (SF-12) Health Survey | 24 weeks
  The SF-12 is a standardized, self-administered questionnaire designed to assess overall health-related quality of life. It includes 12 items that measure physical and mental health components, generating Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. Scores are standardized on a scale where higher values indicate better health status. Both PCS and MCS scores typically range from 0 to 100, with 0 indicating the poorest health and 100 indicating the best possible health status.
Physical Function Measure: Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue and Physical Function Domains | 24 weeks
  The PROMIS is a standardized set of self-reported questionnaires designed to measure health domains. This study includes the fatigue and physical function domains, which assess the participant's perceived level of tiredness and ability to perform daily physical activities. Responses generate standardized T-scores, calibrated to the general population. Higher fatigue T-scores indicate greater fatigue severity.
Aging Biomarkers: Cellular Senescence Markers in Plasma | 24 weeks
  Cellular senescence markers are measured in plasma samples to assess biological aging and cellular stress. These markers may include proteins associated with the senescence-associated secretory phenotype (SASP). Quantification is performed using immunoassays. Higher levels of senescence markers indicate increased cellular senescence.
Difference between biological and chronological age | 24 weeks
  Epigenetic clocks estimate biological age by analyzing DNA methylation patterns at specific CpG sites across the genome. Biological age estimates are compared to chronological age to assess aging acceleration or deceleration. Biological age greater than chronological age indicates accelerated biological aging and potential increased risk of morbidity and mortality. Primary measure is the difference (ΔAge) between biological and chronological ages = reported in years.
Vascular Function Assessment: Reactive Hyperemia Index (RHI) using EndoPAT | 24 weeks
  The RHI is measured using the EndoPAT device, which assesses endothelial function by evaluating changes in digital pulse volume during reactive hyperemia. This non-invasive test involves occluding blood flow in one arm followed by release to induce vasodilation, with pulse amplitude recorded via finger probes. Lower RHI values suggest endothelial dysfunction and increased cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Maria D. Hurtado Andrade, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials